CLINICAL TRIAL: NCT07152808
Title: Clinical Pilot Study to Provide Research Data for TONOREF III Tested to ANSI Z80.10-2014
Brief Title: Clinical Study for TONOREF III Tested to ANSI Z80.10-2014
Status: Completed | Type: Interventional
Sponsor: Nidek Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIDEK-TONOREF-PILOT-0002
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Intraocular Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- TONOREF III and Goldmann Tonometer Measurements (Experimental): Subjects will undergo IOP measurements using both the investigational device (TONOREF III) and the predicate device (Goldmann Applanation Tonometer).
  Interventions: Device: NIDEK TONOREF III; Device: Haag-Streit Goldmann Manual Tonometer

INTERVENTIONS:
Device: NIDEK TONOREF III — The auto ref/kerato/tono/pachymeter TONOREF III is a medical device which measures objective refractive errors, corneal curvature radius, intraocular pressure and corneal thickness of the patient's eye.
Device: Haag-Streit Goldmann Manual Tonometer — Haag-Streit Goldmann Manual Tonometer measures intraocular pressure to aid in the screening and diagnosis of glaucoma

SUMMARY:
The primary objective of this clinical study was to show that tonometry values for TONOREF III, as the representative device of the NIDEK tonometer series, were comparable to the predicate device.

The secondary objective was to demonstrate that the test device was as safe as the predicate device.

ELIGIBILITY:
Inclusion Criteria:

Each subject had to have:

1. been at least 22 years of age of either sex and any race or ethnicity;
2. been willing and able to provide written informed consent prior to any study procedures being performed;
3. been willing and able to follow all instructions and attend all study visits;
4. corneal astigmatism of ≤3D and corneal thickness of 500-600 μm in at least one eye.

Exclusion Criteria:

Each subject had to not to :

1. have only one functional eye;
2. have poor or eccentric fixation in the study eye;
3. have corneal scarring or have had corneal surgery, including corneal laser surgery in the study eye
4. have microphthalmos in the study eye;
5. have buphthalmos in the study eye;
6. be a contact lens wearer in the study eye;
7. have dry eyes;
8. be a lid squeezer - blepharospasm;
9. have nystagmus in the study eye;
10. have keratoconus in the study eye;
11. have any other corneal or conjunctival pathology or infection in the study eye;
12. use medication that affect IOP;
13. current participation in other clinical trials;
14. have a condition or a situation, which in the Investigator's opinion, may put the subject at increased risk, confound study data, or interfere significantly with the subject's study participation.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-02 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TONOREF III and Goldmann Tonometer Measurements
Started | 52
Completed | 42
Not Completed | 10
Not completed — screening failure | 10

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Arm/Group | TONOREF III and Goldmann Tonometer Measurements
Number analyzed (Participants) | 42
Number analyzed (eyes) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 37
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Agreement of Intraocular Pressure
Description: Agreement of the measured IOP between the test device and the predicate device (GAT) for the tonometer function of the TONOREF III. (Agreement means the similarity of results when measurements from the test device and the predicate device are compared against each other.)
Time Frame: 1-2 study visits per subject over the course of 8 days
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | TONOREF III and Goldmann Tonometer Measurements
Number analyzed (Participants) | 42
Number analyzed (eyes) | 80
mmHg
  NIDEK TONOREF III | 18.4 (4.50)
  Haag-Streit GAT | 18.3 (5.11)

2. Secondary Outcome: The Numbers of Adverse Events
Description: To demonstrate that the test device is as safe as GAT
Time Frame: 1-2 study visits per subject over the course of 8 days
Population: No subject had an AE.
Measure: Number; unit: Number of Adverse Event
Arm/Group | TONOREF III and Goldmann Tonometer Measurements
Number analyzed (Participants) | 52
Number of Adverse Event | 0

ADVERSE EVENTS:
Time Frame: 1 to 8 days
Arm/Group | TONOREF III and Goldmann Tonometer Measurements
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 0/52
Other Adverse Events (participants affected / at risk) | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT07152808/Prot_SAP_000.pdf